CLINICAL TRIAL: NCT03471403
Title: Cold Snare Polypectomy for Duodenal Adenomas in Familial Adenomatous Polyposis
Acronym: COPDA
Status: Recruiting | Type: Observational
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Professor Michael Bourke, Director of Gastrointestinal Endoscopy, Western Sydney Local Health District
Other Study IDs: HREC/17/WMEAD/20(5002)
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Familial Adenomatous Polyposis
Keywords: Cold snare polypectomy
MeSH Terms: conditions — Adenomatous Polyposis Coli

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FAP: FAP patients with duodenal adenomas

SUMMARY:
The purpose of this study is to collect prospective observational data regarding patients with diagnosed Familial Adenomatous Polyposis (FAP) undergoing cold snare polypectomy for duodenal adenomas

DETAILED DESCRIPTION:
Familial adenomatous polyposis (FAP) is a autosomal dominant disorder, secondary to a germ-line mutation in the tumour suppressor gene and characterised by multiple colorectal polyps (>100). Typically colorectal adenomas develop in the second and third decade of life. As a result these patients require an endoscopic colonic surveillance program, especially for at-risk family members, which usually begins in the 2nd decade of life starting with annual flexible sigmoidoscopies. The lifetime risk of colorectal cancer (CRC) is 100 percent, if left untreated and patient usually develop CRC in the 4th-5th decade of life. The patient's thus usually progress to a total colectomy.

FAP is also associated with adenomas in the upper gastrointestinal tract and is in nearly 90% of patients with FAP by age 70.Upper gastrointestinal tract screening with gastroscopies commences usually from 25-30 years of age. Usually a duodenoscopy is performed simultaneously to assess for ampullary adenomas. Although surgical procedures have been shown to be effective and have changed the natural history of colorectal cancer in FAP the management of duodenal adenomatosis remains a challenge. The prevalence of FAP associated duodenal adenomas has led to the development of Spigelman classification which assigns surveillance intervals by dividing patient's into four group based on size, histology and severity of dysplasia on histology7. Local endoscopic therapy options available for duodenal adenomatosis include; snare polypectomy, thermal ablation (using a mono/bipolar current) and laser coagulation each with their own limitation. Endoscopic intervention is usually recommended for Spigelman stage II and III disease.

Duodenal endoscopic mucosal resection (EMR) has been shown to be safe and effective methods in removing flat duodenal adenomas in FAP as observed in small case series. However as with colonic EMR these patient's automatically are placed in a higher risk group with the feared complications of delayed bleeding (per and post procedure) and perforation, with the former being as high as 10-15%. The bleeding risk is especially increased in the duodenum due to the rich vascularity of the sub-mucosal layer.

Cold snare polypectomy (CSP) has been shown to be a safe and effective method for removing diminutive colorectal polyps (<8mm) as compared to conventional polypectomy/endoscopic mucosal resection (EMR).

A small case series published the use of a hybrid technique, for duodenal adenomas, where a submucosal injection is performed underneath the lesion to separate the mucosa from the larger sub-mucosal vessels from which bleeding risk is thought to arise. By then performing cold snare piece-meal polypectomy and avoiding the need for thermal therapy risk of delayed bleeding associated is significantly reduced as compared to conventional EMR.

Isolated case report using CSP in non-ampullary duodenal adenomas have shown this technique to be effective.

No large studies to date have examined the use of this technique for duodenal adenomas.

ELIGIBILITY:
Inclusion Criteria:

* Patient's diagnosed with a confirmed diagnosis of FAP (genetic testing) and able to give informed consent to involvement in trial. For patients who do not speak English, an interpreter will be asked to translate the informed consent
* Patients already commenced on endoscopic surveillance for FAP.

Exclusion Criteria:

* Patient's with known strictures/stenosis
* Pregnancy
* Patients who did not consent to study
* Bleeding diathesis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed Familial Adenomatous Polyposis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2027-10-10 (Estimated); Study Completion 2028-10-10 (Estimated)

PRIMARY OUTCOMES:
Number of serious and non-serious adverse events | Three years
  * bleeding risk
  * adenoma recurrence

SECONDARY OUTCOMES:
Duration of endoscopic procedure | Three years
Perforation (peri-procedure and delayed) | Three years
Pain post procedure | Three years
  Measured with 0 - 10 scale
Hospital readmission | Three years
Change in Spigelman stage | Three years

CONTACTS AND LOCATIONS:
Locations (1):
- Westmead Endoscopy Unit, Westmead, New South Wales, Australia